CLINICAL TRIAL: NCT06234306
Title: Molecularly Redefining Small Bowel Adenocarcinoma to Accelerate Precision Patient Care
Acronym: SBAMOL
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Dan Hogdall, MD PhD, Copenhagen University Hospital at Herlev
Other Study IDs: 2312342
Record Dates: First submitted 2024-01-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Small Bowel Adenocarcinoma
Keywords: Small bowel adenocarcinoma; messenger RNA; DNA; T-cell receptor sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-Fixed, Paraffin-Embedded or fresh frozen tissue for DNA, RNA and geospatial analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Small bowel adenocarcinoma is a rare malignancy, and there is limited knowledge about its optimal clinical management and molecular background. The SBAMOL study is an observational biomarker study that aims to identify prognostic and predictive biomarkers. This effort is intended to lay the groundwork for personalized medicine tailored to this specific patient group.

DETAILED DESCRIPTION:
Small bowel adenocarcinoma (SBA), an orphan cancer, has annual diagnoses of 12,070 in the USA and 100 in Denmark. Despite its rarity, patient management should prioritize evidence-based care, but large trials are not feasible, leading to data scarcity and suboptimal care. As a result, SBA is treated like colorectal cancer, yet its prognosis is worse, indicating this parallel approach is insufficient. The grasp on SBAs molecular landscape is limited compared to prevalent cancers. Scant mutational profiling studies, suggest SBA is a heterogeneous disease where subsets resemble other gastrointestinal cancers. This underscores the potential for personalized treatments, including targeted therapies and immunotherapies. Comprehensive molecular characterization, using DNA, RNA, and T-cell receptor characteristics, can provide much-needed strategic direction for patient care and future trials. Capitalizing on this, the investigators propose a comprehensive molecular characterization aiming to develop consensus molecular subtypes that can direct future trials and SBA therapeutic strategies.

The investigators hypothesize that a consensus molecular profiling approach can identify subgroups of SBA with distinct molecular, cellular, and histological characteristics, that will benefit from tailored treatment strategies using chemotherapy, targeted therapy, and immunotherapy.

To explore this hypothesis, the investigators will: (WP1) perform molecular and immunological characterization of tumor tissues from SBA patients (n=200) to establish consensus molecular subtypes of SBA and define their biological attributes; (WP2) ascertain therapeutic avenues tailored to each subtype and devise a molecular algorithm to prospectively categorize individual tumors in real-time, laying the groundwork for molecularly-driven management.

ELIGIBILITY:
Inclusion criteria:

Patients with histologically verified small bowel adenocarcinoma Patients older than 18 years

Exclusion criteria:

Insufficient material for molecular testing Patients registered in Vævsanvendelsesregistret&

Vævsanvendelsesregistret; refers to a central Danish registry where patients can opt out of allowing their biological material to be used for purposes other than their own disease management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with small bowel adenocarcinoma referred to management at participating centers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular characterization of patients with SBA using high-throughput DNA-, mRNA- and T-cell receptor sequencing and targeted protein expression analyses. | 5 years
  Due to the scarce knowledge of the biological background of SBA. The primary endpoint of the study is to present a comprehensive descriptive molecular characterisation of patients with SBA.

SECONDARY OUTCOMES:
Prognostic and predictive DNA biomarkers in patients with SBA | 5 years
  DNA aberrations will associated with disease free, progression free and overall survival. Analysis will be performed using the Oncomine comprehensive plus gene panel. Potential aberrations indicative of targeted treatments will be explored and reported.
Prognostic and predictive mRNA biomarkers in patients with SBA | 5 years
  mRNA aberrations will associated with disease free, progression free and overall survival. Analysis will be performed using high-throughput sequencing. Potential aberrations indicative of targeted treatments will be explored and reported.
Prognostic t-cell receptor biomarkers in patients with SBA | 5 years
  T-cell receptor clonality and diversity will associated with disease free, progression free and overall survival. Analysis will be performed using a high-throughput t-cell receptor sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Høgdall, MD PhD, Principal Investigator — Department of Oncology, Copenhagen University Hospital - Herlev and Gentofte
Locations (3):
- Denmark (3):
  - Department of Oncology, Aarhus University Hospital, Aarhus N
  - Department Surgical Gastroenterology, Copenhagen University Hospital - Rigshospitalet, Copenhagen Ø
  - Department of Oncology Copenhagen University Hospital - Herlev and Gentofte, Herlev

IPD SHARING:
Plan to Share IPD: Undecided
Due to Danish ethical regulations, data can only be shared upon appropriate ethical amendment

REFERENCES:
- [Derived] Dossing RH, Broman JJA, O'Rourke CJ, Tabaksblat EM, Andersen JB, Hansen CP, Poulsen TS, Hogdall EVS, Schou JHV, Hogdall D. Molecularly redefining small bowel adenocarcinoma to accelerate precision patient care - protocol of a multicenter observational cohort biomarker study. BMC Cancer. 2025 Jan 7;25(1):22. doi: 10.1186/s12885-024-13369-1. PMID 39773121